CLINICAL TRIAL: NCT03574610
Title: Supraspinal Mechanisms Involved in Voiding Dysfunction.
Brief Title: Brain Targets in Patients With Bladder Emptying Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, Houston Methodist Hospital Urologist and Research Director, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019329; K12DK083014 (NIH); K23DK118209 (NIH)
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Neurogenic Bladder; Multiple Sclerosis; Voiding Dysfunction
Keywords: Neurogenic bladder; Functional Neuroimaging; Transcranial Rotating Permanent Magnet Stimulator (TRPMS)
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects with Multiple Sclerosis and Voiding Dysfunction (Experimental): Subjects with Multiple Sclerosis (MS) and voiding dysfunction (VD). In this group 'Transcranial Rotating Permanent Magnet Stimulator (TRPMS)' device will be used.
  Interventions: Device: Transcranial Rotating Permanent Magnet Stimulator (TRPMS)

INTERVENTIONS:
Device: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) — TRPMS is a wearable non-invasive transcranial rotating permanent magnet stimulator. It has been determined to be a Non Significant Risk device by the FDA.
  The amount and frequency of therapy are prescribed by the physician, and the device is custom configured to the patient to deliver the required amount of treatment. The device does not turn on until it is time for the treatment. It consists of three main parts: Neoprene cap with microstimulator(s), stimulator console (device controller box) and the tablet with TRPMS app which activates the console. The neoprene cap prevents the microstimulator(s) from coming in direct contact with the scalp. Microstimulators deliver the magnetic stimulation to the brain based on a prescription program uploaded in the stimulator controller.

SUMMARY:
The goal of this study is to identify brain centers specifically associated with "initiation of voiding" in patients with neurogenic bladder dysfunction. Currently there is no study that has evaluated brain centers involved in initiation of voiding in patients with neurogenic voiding dysfunction.

Patients with neurogenic bladder secondary to etiologies such as Multiple Sclerosis, Parkinson's disease, and Cerebrovascular accidents will be recruited in this study. Patients will be categorized into 2 groups, those who have trouble emptying their bladder and those who urinate appropriately. Our existing and unique functional magnetic resonance imaging (fMRI)/ urodynamics (UDS) platform is an ideal platform to identify brain regions involved in bladder emptying disorders as seen in patients with neurogenic bladder dysfunction and will be used for this study. After characterizing brain regions involved in bladder emptying, the investigator propose to use noninvasive transcutaneous magnetic stimulation in a subset of patients with voiding dysfunction in aim 3.

DETAILED DESCRIPTION:
Difficulty in bladder emptying (Voiding dysfunction,VD) is a costly urinary condition that leads to urinary tract infections/stones, sepsis, bladder loss, and permanent kidney damage. VD can be present in patients with or without neurologic/brain disorders. Currently the only available therapies for VD include bladder catheters or intermittent self-catheterization. Catheterization is a burden especially in patients with nerve damage, hand skills may be limited. The cost and morbid side effects of catheterizations in patients (blood in the urine, pain, trauma, strictures, and infections) requires investigators to develop new therapies that are beyond the bladder. Such new therapies could target the brain (where bladder control is located).

In this proposal, investigators plan to further characterize the brain regions involved in bladder emptying for each patient and ,perform brain modulation, targeting these regions as a possible therapy for VD.

Patients with bladder dysfunction will be divided into two groups: Group 1: patients with VD; and Group 2: patients without VD. Specific Aim 1: To evaluate brain pattern in both groups and compare them to each other at the time of bladder emptying. Specific Aim 2: To evaluate reliability of the nerve fibers in the brain and see whether damage to these fibers is related to difficulty emptying the bladder. Specific Aim 3: To perform non-invasive brain stimulation on specific regions of the brain responsible for bladder control to improve bladder emptying.

This study is an interventional Study: The investigators have completed a well-powered study on twenty-seven female MS patients during their bladder storage phase. Aims 1 and 2 use the data from previously completed trial and investigators will perform additional imaging analysis on it. Aim 3 is a new and small trial in which investigators planned to modulate the regions of the brain that are related to bladder control.

Approximately 16 study participants will be enrolled at Houston Methodist, and 16 throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for subjects with neurogenic bladder:

* Patients with clinical diagnosis of neurogenic bladder
* History of any neurologic illness or injury (including but not limited to spinal cord injury, Multiple Sclerosis, Stroke, spina bifida, Parkinson's, major spine surgery)
* 18 years or older

Specifics for MS patients:

Adult female patients with clinically stable MS [Expanded Disability Status Score (EDSS) ≤6.5], with bladder symptoms ≥3 months, will be screened. Patients will be considered to have VD if they have an increased Postvoid Residual (≥ 20% Maximum Cystometric Capacity). Patients who perform self-catheterization will be included in the VD category as well.

Exclusion Criteria:

Exclusion Criteria for subjects with neurogenic bladder:

* Men (for aims 1 and 2 only), anatomical bladder outlet obstruction (anti-incontinence procedures, urethral strictures, or advanced pelvic organ prolapse). Severe debilitating MS, history of seizures, pregnancy or planning to become pregnant, contraindications to MRI, history of augmentation cystoplasty. Patients with active urinary tract infection (UTI) can be treated and subsequently screened for the trial.
* Positive urine pregnancy test at enrollment (There are no known risks to a subject's fetus. There is no known teratogenic risk associated with urodynamics or fMRI) - Cognitively impaired patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panicker JN, Fowler CJ, Kessler TM. Lower urinary tract dysfunction in the neurological patient: clinical assessment and management. Lancet Neurol. 2015 Jul;14(7):720-32. doi: 10.1016/S1474-4422(15)00070-8. PMID 26067125
- [Background] Kuhtz-Buschbeck JP, Gilster R, van der Horst C, Hamann M, Wolff S, Jansen O. Control of bladder sensations: an fMRI study of brain activity and effective connectivity. Neuroimage. 2009 Aug 1;47(1):18-27. doi: 10.1016/j.neuroimage.2009.04.020. Epub 2009 Apr 14. PMID 19371782
- [Background] Shy M, Fung S, Boone TB, Karmonik C, Fletcher SG, Khavari R. Functional magnetic resonance imaging during urodynamic testing identifies brain structures initiating micturition. J Urol. 2014 Oct;192(4):1149-54. doi: 10.1016/j.juro.2014.04.090. Epub 2014 Apr 21. PMID 24769029
- [Background] Khavari R, Karmonik C, Shy M, Fletcher S, Boone T. Functional Magnetic Resonance Imaging with Concurrent Urodynamic Testing Identifies Brain Structures Involved in Micturition Cycle in Patients with Multiple Sclerosis. J Urol. 2017 Feb;197(2):438-444. doi: 10.1016/j.juro.2016.09.077. Epub 2016 Sep 21. PMID 27664581
- [Background] Kuhtz-Buschbeck JP, van der Horst C, Wolff S, Filippow N, Nabavi A, Jansen O, Braun PM. Activation of the supplementary motor area (SMA) during voluntary pelvic floor muscle contractions--an fMRI study. Neuroimage. 2007 Apr 1;35(2):449-57. doi: 10.1016/j.neuroimage.2006.12.032. Epub 2007 Jan 9. PMID 17293127
- [Background] Kuhtz-Buschbeck JP, van der Horst C, Pott C, Wolff S, Nabavi A, Jansen O, Junemann KP. Cortical representation of the urge to void: a functional magnetic resonance imaging study. J Urol. 2005 Oct;174(4 Pt 1):1477-81. doi: 10.1097/01.ju.0000173007.84102.7c. PMID 16145475
- [Background] Blok BF, Sturms LM, Holstege G. Brain activation during micturition in women. Brain. 1998 Nov;121 ( Pt 11):2033-42. doi: 10.1093/brain/121.11.2033. PMID 9827764
- [Background] Blok BF, Willemsen AT, Holstege G. A PET study on brain control of micturition in humans. Brain. 1997 Jan;120 ( Pt 1):111-21. doi: 10.1093/brain/120.1.111. PMID 9055802
- [Background] Centonze D, Petta F, Versace V, Rossi S, Torelli F, Prosperetti C, Rossi S, Marfia GA, Bernardi G, Koch G, Miano R, Boffa L, Finazzi-Agro E. Effects of motor cortex rTMS on lower urinary tract dysfunction in multiple sclerosis. Mult Scler. 2007 Mar;13(2):269-71. doi: 10.1177/1352458506070729. Epub 2007 Jan 29. PMID 17439897
- [Background] Choksi D, Schott B, Tran K, Jang R, Hasan KM, Lincoln JA, Jalali A, Karmonik C, Salazar B, Khavari R. Disruption of specific white matter tracts is associated with neurogenic lower urinary tract dysfunction in women with multiple sclerosis. Neurourol Urodyn. 2023 Jan;42(1):239-248. doi: 10.1002/nau.25075. Epub 2022 Nov 2. PMID 36321777
- [Result] Khavari R, Tran K, Helekar SA, Shi Z, Karmonik C, Rajab H, John B, Jalali A, Boone T. Noninvasive, Individualized Cortical Modulation Using Transcranial Rotating Permanent Magnet Stimulator for Voiding Dysfunction in Women with Multiple Sclerosis: A Pilot Trial. J Urol. 2022 Mar;207(3):657-668. doi: 10.1097/JU.0000000000002297. Epub 2021 Oct 25. PMID 34694911
- [Result] Jang Y, Tran K, Shi Z, Christof K, Choksi D, Salazar BH, Lincoln JA, Khavari R. Predictors for outcomes of noninvasive, individualized transcranial magnetic neuromodulation in multiple sclerosis women with neurogenic voiding dysfunction. Continence (Amst). 2022 Dec;4:100517. doi: 10.1016/j.cont.2022.100517. Epub 2022 Oct 19. PMID 36568960
- [Result] Shi Z, Karmonik C, Soltes A, Tran K, Lincoln JA, Boone T, Khavari R. Altered bladder-related brain network in multiple sclerosis women with voiding dysfunction. Neurourol Urodyn. 2022 Sep;41(7):1612-1619. doi: 10.1002/nau.25008. Epub 2022 Jul 17. PMID 35842826
- [Derived] Tran K, Shi Z, Karmonik C, John B, Rajab H, Helekar SA, Boone T, Khavari R. Therapeutic effects of non-invasive, individualized, transcranial neuromodulation treatment for voiding dysfunction in multiple sclerosis patients: study protocol for a pilot clinical trial. Pilot Feasibility Stud. 2021 Mar 24;7(1):83. doi: 10.1186/s40814-021-00825-z. PMID 33757581

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Multiple Sclerosis and Voiding Dysfunction: Subjects with Multiple Sclerosis (MS) and voiding dysfunction (VD). In this group 'Transcranial Rotating Permanent Magnet Stimulator (TRPMS)' device will be used.
  Transcranial Rotating Permanent Magnet Stimulator (TRPMS): TRPMS is a wearable non-invasive transcranial rotating permanent magnet stimulator. It has been determined to be a Non Significant Risk device by the FDA.
  The amount and frequency of therapy are prescribed by the physician, and the device is custom configured to the patient to deliver the required amount of treatment. The device does not turn on until it is time for the treatment. It consists of three main parts: Neoprene cap with microstimulator(s), stimulator console (device controller box) and the tablet with TRPMS app which activates the console. The neoprene cap prevents the microstimulator(s) from coming in direct contact with the scalp. Microstimulators deliver the magnetic stimulation to the brain based on a prescription program uploaded in the stimulator controller.
Period: Overall Study
Arm/Group | Subjects With Multiple Sclerosis and Voiding Dysfunction
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Multiple Sclerosis and Voiding Dysfunction
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 53.40 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Number of participants [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Activity After Treatment Measured Using Functional MRI
Description: Here we measured changes in brain activation in modulated brain regions of interest (ROI) via blood oxygen level-dependent (BOLD) signals during "strong desire to void" and "voiding initiation (attempt)". We determined if there was a significant increase or decrease in activity (voxel signal) after treatment using the following criteria: 1) increase in activation was defined as T-value greater than 2.074 and 2) decrease in activation was defined as T-value less than 2.074.
Time Frame: Baseline to three weeks
Population: Eleven patients were eligible and consented to participate. One withdrew before baseline scan, and 10 received the treatment and completed all their scans and assessments (July 2019 - December 2020) and were included in the analysis. Amongst 8 patients who completed their 4-month follow-ups, 1 could not return for an in-person visit and only her validated questionnaires were collected.
Measure: Mean (Full Range); unit: BOLD fMRI T-Value
Groups:
- Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis: Transcranial Rotating Permanent Magnet Stimulator (TRPMS): TRPMS is a wearable non-invasive transcranial rotating permanent magnet stimulator. It has been determined to be a Non Significant Risk device by the FDA.
  The amount and frequency of therapy are prescribed by the physician, and the device is custom configured to the patient to deliver the required amount of treatment. The device does not turn on until it is time for the treatment. It consists of three main parts: Neoprene cap with microstimulator(s), stimulator console (device controller box) and the tablet with TRPMS app which activates the console. The neoprene cap prevents the microstimulator(s) from coming in direct contact with the scalp. Microstimulators deliver the magnetic stimulation to the brain based on a prescription program uploaded in the stimulator controller.
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
BOLD fMRI T-Value
  Strong desire to void: L inferior frontal gyrus | 2.759234 [-6.306071 to 5.683107]
  Strong desire to void: L superior temporal gyrus | 3.423569 [-6.306071 to 5.683107]
  Strong desire to void: L inferior temporal gyrus | 3.000987 [-6.306071 to 5.683107]
  Strong desire to void: L middle temporal gyrus | 3.094914 [-6.306071 to 5.683107]
  Strong desire to void: R middle temporal gyrus | 4.046153 [-6.306071 to 5.683107]
  Strong desire to void: L inferior parietal lobule | 2.950705 [-6.306071 to 5.683107]
  Strong desire to void: R inferior parietal lobule | 4.215242 [-6.306071 to 5.683107]
  Strong desire to void: R paracentral lobule | 2.799833 [-6.306071 to 5.683107]
  Strong desire to void: R superior parietal lobule | 4.003400 [-6.306071 to 5.683107]
  Strong Desire to void: R supplementary motor area | 4.317012 [-6.306071 to 5.683107]
  Strong Desire to void: L postcentral gyrus | 5.520249 [-6.306071 to 5.683107]
  Strong Desire to void: R postcentral gyrus | 5.455663 [-6.306071 to 5.683107]
  Strong Desire to void: L angular gyrus | 3.369907 [-6.306071 to 5.683107]
  Strong Desire to void: R supramarginal gyrus | 4.578173 [-6.306071 to 5.683107]
  Strong Desire to void: L superior medial gyrus | 3.745239 [-6.306071 to 5.683107]
  Strong Desire to void: L inferior occipital gyrus | 5.683107 [-6.306071 to 5.683107]
  Strong Desire to void: L middle cingulate cortex | 3.782596 [-6.306071 to 5.683107]
  Strong Desire to void: R middle cingulate cortex | 3.693368 [-6.306071 to 5.683107]
  Strong Desire to void: R posterior cingulate cortex | 3.913861 [-6.306071 to 5.683107]
  Strong Desire to void: L thalamus | 2.753587 [-6.306071 to 5.683107]
  Strong Desire to void: R thalamus | 3.373487 [-6.306071 to 5.683107]
  Strong Desire to void: L precuneus | 4.345939 [-6.306071 to 5.683107]
  Strong Desire to void: R precuneus | 3.767377 [-6.306071 to 5.683107]
  Strong Desire to void: L caudate nucleus | 4.684247 [-6.306071 to 5.683107]
  Strong Desire to void: L hippocampus | 3.027731 [-6.306071 to 5.683107]
  Strong Desire to void: L putamen | 3.695211 [-6.306071 to 5.683107]
  Strong Desire to void: L precentral gyrus | -3.990877 [-6.306071 to 5.683107]
  Strong Desire to void: R precentral gyrus | -4.272436 [-6.306071 to 5.683107]
  Strong Desire to void: L insula lobe | -2.769022 [-6.306071 to 5.683107]
  Strong Desire to void: L superior frontal gyrus | -3.345682 [-6.306071 to 5.683107]
  Strong Desire to void: L middle frontal gyrus | -2.921264 [-6.306071 to 5.683107]
  Strong Desire to void: R cerebellum | -3.007422 [-6.306071 to 5.683107]
  Strong Desire to void: R fusiform gyrus | -6.306071 [-6.306071 to 5.683107]
  Voiding initiation: L postcentral gyrus | 4.999096 [-6.306071 to 5.683107]
  Voiding initiation: R postcentral gyrus | 4.028872 [-6.306071 to 5.683107]
  Voiding initiation: L precentral gyrus | 4.425272 [-6.306071 to 5.683107]
  Voiding initiation: R precentral gyrus | 4.393749 [-6.306071 to 5.683107]
  Voiding initiation: L superior temporal gyrus | 3.324719 [-6.306071 to 5.683107]
  Voiding initiation: R superior temporal gyrus | 3.313340 [-6.306071 to 5.683107]
  Voiding initiation: L middle temporal gyrus | 4.935463 [-6.306071 to 5.683107]
  Voiding initiation: R middle temporal gyrus | 5.257658 [-6.306071 to 5.683107]
  Voiding initiation: L inferior temporal gyrus | 4.281283 [-6.306071 to 5.683107]
  Voiding initiation: L supramarginal gyrus | 3.906453 [-6.306071 to 5.683107]
  Voiding initiation: R supramarginal gyrus | 5.236864 [-6.306071 to 5.683107]
  Voiding initiation: L inferior occipital gyrus | 3.065269 [-6.306071 to 5.683107]
  Voiding initiation: R superior occipital gyrus | 4.129290 [-6.306071 to 5.683107]
  Voiding initiation: R middle occipital gyrus | 4.078387 [-6.306071 to 5.683107]
  Voiding initiation: L inferior frontal gyrus (p. Orbitalis) | 4.038723 [-6.306071 to 5.683107]
  Voiding initiation: L inferior frontal gyrus (p. Triangularis) | 4.274477 [-6.306071 to 5.683107]
  Voiding initiation: L inferior frontal gyrus (p. Opercularis) | 2.819778 [-6.306071 to 5.683107]
  Voiding initiation: R inferior frontal gyrus (p. Orbitalis) | 3.072036 [-6.306071 to 5.683107]
  Voiding initiation: R inferior frontal gyrus (p. Triangularis) | 3.645947 [-6.306071 to 5.683107]
  Voiding initiation: L cerebellum | 4.210466 [-6.306071 to 5.683107]
  Voiding initiation: L rectal gyrus | 4.637410 [-6.306071 to 5.683107]
  Voiding initiation: R rectal gyrus | 3.535679 [-6.306071 to 5.683107]
  Voiding initiation: L superior medial gyrus | 3.402534 [-6.306071 to 5.683107]
  Voiding initiation: R superior medial gyrus | 3.136795 [-6.306071 to 5.683107]
  Voiding initiation: L superior frontal gyrus | 2.455777 [-6.306071 to 5.683107]
  Voiding initiation: R superior frontal gyrus | 3.053638 [-6.306071 to 5.683107]
  Voiding initiation: L middle frontal gyrus | 3.798942 [-6.306071 to 5.683107]
  Voiding initiation: R middle frontal gyrus | 3.897008 [-6.306071 to 5.683107]
  Voiding initiation: L supplementary motor area | 2.518869 [-6.306071 to 5.683107]
  Voiding initiation: R supplementary motor area | 4.614616 [-6.306071 to 5.683107]
  Voiding initiation: L paracentral lobule | 3.324731 [-6.306071 to 5.683107]
  Voiding initiation: R paracentral lobule | 5.114769 [-6.306071 to 5.683107]
  Voiding initiation: R superior parietal lobule | 4.184497 [-6.306071 to 5.683107]
  Voiding initiation: R inferior parietal lobule | 4.545515 [-6.306071 to 5.683107]
  Voiding initiation: L superior orbital gyrus | 3.721826 [-6.306071 to 5.683107]
  Voiding initiation: L middle orbital gyrus | 5.286532 [-6.306071 to 5.683107]
  Voiding initiation: R middle orbital gyrus | 3.078467 [-6.306071 to 5.683107]
  Voiding initiation: R calcarine gyrus | 3.512251 [-6.306071 to 5.683107]
  Voiding initiation: L calcarine gyrus | 3.551130 [-6.306071 to 5.683107]
  Voiding initiation: L anterior cingulate cortex | 4.160711 [-6.306071 to 5.683107]
  Voiding initiation: L middle cingulate cortex | 3.181774 [-6.306071 to 5.683107]
  Voiding initiation: R middle cingulate cortex | 3.946584 [-6.306071 to 5.683107]
  Voiding initiation: R angular gyrus | 4.111778 [-6.306071 to 5.683107]
  Voiding initiation: L thalamus | 3.140146 [-6.306071 to 5.683107]
  Voiding initiation: R thalamus | 3.255678 [-6.306071 to 5.683107]
  Voiding initiation: L precuneus | 4.921595 [-6.306071 to 5.683107]
  Voiding initiation: R precuneus | 4.093221 [-6.306071 to 5.683107]
  Voiding initiation: R caudate nucleus | 3.857368 [-6.306071 to 5.683107]
  Voiding initiation: L putamen | 3.188081 [-6.306071 to 5.683107]
  Voiding initiation: L amygdala | 2.479540 [-6.306071 to 5.683107]
  Voiding initiation: R insula lobe | 3.000530 [-6.306071 to 5.683107]
  Voiding initiation: L rolandic operculum | 2.860924 [-6.306071 to 5.683107]
  Voiding initiation: L hippocampus | -4.078490 [-6.306071 to 5.683107]
  Voiding initiation: R hippocampus | -3.109341 [-6.306071 to 5.683107]
  Voiding initiation: R fusiform gyrus | -3.328545 [-6.306071 to 5.683107]
  Voiding initiation: R rolandic operculum | -3.971051 [-6.306071 to 5.683107]
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L inferior frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Desire to void: L superior temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 3: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L inferior temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 4: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L middle temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 5: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R middle temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 6: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L inferior parietal lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 7: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R inferior parietal lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 8: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R paracentral lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 9: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R superior parietal lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 10: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R supplementary motor area; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 11: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L postcentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 12: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R postcentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 13: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L angular gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 14: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R supramarginal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 15: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L superior medial gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 16: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L inferior occipital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 17: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L middle cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 18: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R middle cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 19: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R posterior cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 20: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L thalamus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 21: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R thalamus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 22: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L precuneus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 23: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R precuneus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 24: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L caudate nucleus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 25: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire void: L hippocampus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 26: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L hippocampus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 27: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L putamen; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 28: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L precentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 29: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R precentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 30: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L insula lobe; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 31: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L superior frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 32: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: L middle frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 33: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R cerebellum; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 34: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Strong desire to void: R fusiform gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 35: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L postcentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 36: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R postcentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 37: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L precentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 38: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R precentral gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 39: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L superior temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 40: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R superior temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 41: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L middle temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 42: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R middle temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 43: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L inferior temporal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 44: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L supramarginal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 45: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R supramarginal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 46: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding Initiation: L inferior occipital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 47: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R superior occipital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 48: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding Initiation: R middle occipital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 49: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L inferior frontal gyrus (p. Orbitalis); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 50: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L inferior frontal gyrus (p. Triangularis); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 51: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L inferior frontal gyrus (p. Opercularis); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 52: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R inferior frontal gyrus (p. Orbitalis); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 53: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R inferior frontal gyrus (p. Triangularis); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 54: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L cerebellum; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 55: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L rectal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 56: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R rectal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 57: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L superior medial gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 58: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R superior medial gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 59: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L superior frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 60: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R superior frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 61: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L middle frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 62: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R middle frontal gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 63: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L supplementary motor area (SMA); Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 64: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R SMA; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 65: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L paracentral lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 66: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R paracentral lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 67: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R superior parietal lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 68: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R inferior parietal lobule; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 69: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L superior orbital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 70: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L middle orbital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 71: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R middle orbital gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 72: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R calcarine gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 73: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L calcarine gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 74: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L anterior cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 75: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L middle cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 76: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R middle cingulate cortex; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 77: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R angular gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 78: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L thalamus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 79: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R thalamus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 80: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L precuneus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 81: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R precuneus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 82: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R caudate nucleus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 83: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L putamen; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 84: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L amygdala; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 85: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R insula lobe; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 86: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L rolandic operculum; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 87: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: L hippocampus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 88: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R hippocampus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 89: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R fusiform gyrus; Test type: Other; p < 0.05, Student's t-test
Statistical Analysis 90: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voiding initiation: R rolandic operculum; Test type: Other; p < 0.05, Student's t-test

2. Secondary Outcome: Changes in Objective Clinical Outcomes Following Treatment
Description: The objective clinical assessment included changes in post void residual (PVR), voided volume (VV) and bladder capacity (BC) in participants after treatment as compared to baseline. PVR measures the volume of urine (cc/mL) that is left after voiding. VV measures the volume of urine that is voided (cc/mL). BC measures the volume of urine (cc/mL) the bladder has a capacity to hold, this value is calculated by adding the VV + PVR values obtained.
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
mL
  Voided volume baseline | 188.1 (112.21)
  Voided volume post-treatment | 218.80 (110.12)
  Voided volume 4 month follow-up: number analyzed (Participants) | 8
  Voided volume 4 month follow-up | 189.88 (106.32)
  PVR baseline | 193.10 (83.46)
  PVR post-treatment | 98.70 (89.37)
  PVR 4 month follow-up: number analyzed (Participants) | 8
  PVR 4 month follow-up | 160.70 (142.93)
  Bladder capacity baseline | 381.20 (152.37)
  Bladder capacity post-treatment | 317.50 (144.11)
  Bladder capacity 4 month follow-up | 350.63 (226.32)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voided volume - baseline vs post-treatment; Test type: Other; p = 0.45, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Voided volume - baseline vs 4 month follow-up; Test type: Other; p = 0.39, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test. (Only used the 8 participants that had data for baseline and 4 month follow-up for statistical calculations)
Statistical Analysis 3: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; PVR - baseline vs post-treatment; Test type: Other; p = 0.014, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 4: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; PVR - baseline vs 4 month follow-up; Test type: Other; p = 0.66, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Bladder capacity - baseline vs post-treatment; Test type: Other; p = 0.31, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 6: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Bladder capacity - baseline vs 4 month follow-up; Test type: Other; p = 0.001, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

3. Secondary Outcome: Changes in %Post-Void Residual/Bladder Capacity (PVR/BC) Following Treatment
Description: Objective clinical assessments included changes in post void residual (PVR) and bladder capacity in participants after treatment. PVR measures the volume of urine (cc/mL) that is left after voiding. BC measures the volume of urine (cc/mL) the bladder has a capacity to hold. % PVR/BC measures how much of the overall volume is left after voiding, showing how efficient a voiding is before and after treatment.
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
Percentage
  %PVR/BC (at baseline) | 54.04 (17.48)
  %PVR/BC (post-treatment) | 29.46 (22.08)
  %PVR/BC (at 4 month follow-up): number analyzed (Participants) | 8
  %PVR/BC (at 4 month follow-up) | 42.08 (18.97)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; % PVR/BC - baseline vs post-treatment; Test type: Other; p = 0.004, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; %PVR/BC - baseline vs 4 month follow-up; Test type: Other; p = 0.038, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

4. Secondary Outcome: Changes in Non-instrumented Uroflow Variable Qmax Following Treatment
Description: The objective clinical assessment included changes in non-instrumented uroflow variables such as Qmax, in participants after treatment as compared to baseline. Qmax values reported here correspond to the peak urine flow (mL/s) seen during uroflowmetry testing.
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
mL/sec
  Qmax at baseline | 22.2 (14.76)
  Qmax post-treatment | 31.00 (15.17)
  Qmax at 4 month follow-up: number analyzed (Participants) | 8
  Qmax at 4 month follow-up | 25.50 (14.25)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Qmax - baseline vs post-treatment; Test type: Other; p = 0.19, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Max - baseline vs 4 month follow-up; Test type: Other; p = 0.91, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

5. Secondary Outcome: Changes in Liverpool Nomogram Following Treatment
Description: The objective clinical assessment included changes in non-instrumented uroflow variables such as Liverpool nomogram in participants after treatment as compared to baseline. The Liverpool nomogram provides normal reference ranges for the maximum and average urine flow rates over a wide range of voided volumes. It is presented as a percentile ranking depending on the flow rate and voided volume for each participant.
Time Frame: Baseline, after treatment and 4 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
Percentile
  Liverpool Nomogram baseline | 34.00 (36.12)
  Liverpool Nomogram post-treatment | 62.80 (32.90)
  Liverpool Nomogram 4 month follow-up: number analyzed (Participants) | 8
  Liverpool Nomogram 4 month follow-up | 49.63 (36.23)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Liverpool nomogram percentile - baseline vs post-treatment; Test type: Other; p = 0.13, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; Liverpool nomogram percentile - baseline vs 4 month follow-up; Test type: Other; p = 0.26, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

6. Secondary Outcome: Changes in Subjective Clinical Outcomes Following Treatment - Urinary Distress Inventory, Short Form (UDI-6) Questionnaire
Description: Our subjective clinical assessment included changes in validated questionnaires. This assessment has 6 questions and is used to assess life quality and symptom distress for urinary incontinence in women. We report raw scores here for questions pertaining to voiding symptoms. Each question has the following score range: 0-4 (with the highest score associated with worse symptoms).
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
Score on a scale
  UDI-6 Q1 baseline | 3.10 (1.45)
  UDI-6 Q1 post-treatment | 2.70 (1.25)
  UDI-6 Q1 4 month follow-up: number analyzed (Participants) | 8
  UDI-6 Q1 4 month follow-up | 1.88 (1.46)
  UDI-6 Q2 baseline | 2.50 (1.51)
  UDI-6 Q2 post-treatment | 2.20 (1.48)
  UDI-6 Q2 4 month follow-up: number analyzed (Participants) | 8
  UDI-6 Q2 4 month follow-up | 1.50 (1.20)
  UDI-6 Q5 baseline | 3.30 (1.06)
  UDI-6 Q5 post-treatment | 2.20 (1.55)
  UDI-6 Q5 4 month follow-up: number analyzed (Participants) | 8
  UDI-6 Q5 4 month follow-up | 1.38 (1.30)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 Q1 - baseline vs post-treatment; Test type: Other; p = 0.40, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 Q1 - baseline vs 4 month follow-up; Test type: Other; p = 0.086, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 Q2 - baseline vs post-treatment; Test type: Other; p = 0.54, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 4: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 Q2 - baseline vs 4 month follow-up; Test type: Other; p = 0.19, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 Q5 - baseline vs post-treatment; Test type: Other; p = 0.04, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 6: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; UDI-6 5 - baseline vs 4 month follow-up; Test type: Other; p = 0.026, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

7. Secondary Outcome: Changes in Subjective Clinical Outcomes Following Treatment - American Urological Association Symptom Score (AUASS) Questionnaire
Description: Our subjective clinical assessment included changes in validated questionnaires. This assessment has 8 questions and is used to assess how bothersome urinary symptoms are and quality of life. We report raw scores here for questions pertaining to voiding symptoms. Questions 1-7 have the following score range: 0-5 (with the highest score associated with worse symptoms). The last question pertains to quality of life and has a score range of: 0-6 (with the highest score associated with very reduced quality of life).
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
Score on a scale
  AUSS Q3 baseline | 4.30 (1.57)
  AUSS Q3 post-treatment | 2.90 (1.52)
  AUSS Q3 4 month follow-up: number analyzed (Participants) | 8
  AUSS Q3 4 month follow-up | 3.00 (1.77)
  AUSS Q5 baseline | 2.60 (1.84)
  AUSS Q5 post-treatment | 2.30 (1.89)
  AUSS Q5 4 month follow-up: number analyzed (Participants) | 8
  AUSS Q5 4 month follow-up | 1.88 (1.73)
  AUSS Q7 baseline | 2.80 (1.14)
  AUSS Q7 post-treatment | 2.20 (0.92)
  AUSS Q7 4 month follow-up: number analyzed (Participants) | 8
  AUSS Q7 4 month follow-up | 2.13 (1.36)
  AUSS Q8 baseline | 4.20 (1.69)
  AUSS Q8 post-treatment | 3.50 (1.35)
  AUSS Q8 4 month follow-up: number analyzed (Participants) | 8
  AUSS Q8 4 month follow-up | 2.75 (1.98)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q3 - baseline vs post-treatment; Test type: Other; p = 0.044, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q3 - baseline vs 4 month follow-up; Test type: Other; p = 0.017, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q5 - baseline vs post-treatment; Test type: Other; p = 0.54, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 4: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q5 - baseline vs 4 month follow-up; Test type: Other; p = 0.503, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q7 - baseline vs post-treatment; Test type: Other; p = 0.023, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 6: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q7 - baseline vs 4 month follow-up; Test type: Other; p = 0.049, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q8 - baseline vs post-treatment; Test type: Other; p = 0.089, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 8: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; AUASS Q8 - baseline vs 4 month follow-up; Test type: Other; p = 0.161, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

8. Secondary Outcome: Changes in Subjective Clinical Outcomes Following Treatment - Neurogenic Bladder Symptom Score (NBSS) Questionnaire
Description: Our subjective clinical assessment included changes in validated questionnaires. This assessment has 24 questions that measure bladder symptoms across 3 different domains: incontinence (score range: 0-29), storage and voiding (score range: 0-22), and consequences (score range: 0-23); the highest score is associated with worse symptoms. The last question focuses on quality of life scored from 0 (pleased) to 4 (unhappy). We report raw scores here for all domains and QoL.
Time Frame: Baseline, after treatment and 4 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis
Number analyzed (Participants) | 10
Score on a scale
  NBSS (Incontinence) baseline | 11.70 (5.91)
  NBSS (Incontinence) post-treatment | 9.00 (6.11)
  NBSS (Incontinence) 4 month follow-up: number analyzed (Participants) | 8
  NBSS (Incontinence) 4 month follow-up | 9.88 (6.15)
  NBSS (Storage and Voiding) baseline | 15.00 (2.62)
  NBSS (Storage and Voiding) post-treatment | 14.10 (2.56)
  NBSS (Storage and Voiding) 4 month follow-up: number analyzed (Participants) | 8
  NBSS (Storage and Voiding) 4 month follow-up | 11.88 (2.17)
  NBSS (Consequences) baseline | 5.00 (2.05)
  NBSS (Consequences) post-treatment | 4.60 (2.50)
  NBSS (Consequences) 4 month follow-up: number analyzed (Participants) | 8
  NBSS (Consequences) 4 month follow-up | 5.63 (1.06)
  NBSS (QoL) baseline | 2.80 (1.32)
  NBSS (QoL) post-treatment | 2.10 (1.10)
  NBSS (QoL) 4 month follow-up: number analyzed (Participants) | 8
  NBSS (QoL) 4 month follow-up | 1.50 (1.31)
Statistical Analysis 1: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Incontinence) - baseline vs post-treatment; Test type: Other; p = 0.010, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 2: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Incontinence) - baseline vs 4 month follow-up; Test type: Other; p = 0.41, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Storage and Voiding) - baseline vs post-treatment; Test type: Other; p = 0.32, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 4: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Storage and Voiding) - baseline vs 4 month follow-up; Test type: Other; p = 0.02, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Consequences) - baseline vs post-treatment; Test type: Other; p = 0.34, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; Paired t-test
Statistical Analysis 6: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (Consequences) - baseline vs 4 month follow-up; Test type: Other; p = 0.61, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (QoL) - baseline vs post-treatment; Test type: Other; p = 0.02, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 8: Comparison: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) in Subjects With Multiple Sclerosis; NBSS (QoL) - baseline vs 4 month follow-up; Test type: Other; p = 0.07, t-test, 2 sided — Threshold for statistical significance used P-value <0.05; [statistical method as in outcome 2, analysis 2]

ADVERSE EVENTS:
Time Frame: Safety was measured by the incidence of patient or investigator-reported adverse events, monitored by the study team and via questionnaires (regarding mood, pain, dizziness, and other sensations) collected at each treatment session. [Time Frame: acute, up to 6 months]
Arm/Group | Subjects With Multiple Sclerosis and Voiding Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
This is a pilot study with a small sample size of 10 women and no controls. Other potential limitations of this study include the supine position during the fMRI/UDS examination, which could pose difficulty for subjects to void in the scanner. MS is a heterogeneous disease, and the observed changes in outcomes could be a result of historical changes unrelated to treatment, or depending on baseline factors such as location of lesion burdens or duration of MS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT03574610/Prot_SAP_001.pdf